CLINICAL TRIAL: NCT04777370
Title: Are There Differences in Range of Motion, Glenohumeral Translation, and Rotator Cuff Activity Following Shoulder Mobilization, Stretching, or Thoracic Manipulation?
Brief Title: Combined Effects of Manual Therapy on the Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hartford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: PRO2021000105
Record Dates: First submitted 2021-02-22; First posted 2021-03-02 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: Range of Motion; Manual Therapies; Shoulder Joint Disorder
Keywords: shoulder; Glenohumeral Internal Rotation Deficit (GIRD); joint play; muscular activity

STUDY DESIGN:
Intervention Model Description: All participants will undergo a single intervention during the first session, and then combined thoracic manipulation and a repeat of the prior intervention at the second session.
Who Masked: Outcomes Assessor
Masking Description: Assessment of electromyographic (EMG) activity, IR ROM pre-post intervention, and glenohumeral translation via ultrasound will be performed by a blinded assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sleeper stretch + thoracic manipulation (Experimental): The group will receive the sleeper stretch at session #1, and a thoracic manipulation followed by the sleeper stretch at session #2.
  Interventions: Other: Sleeper stretch; Other: thoracic manipulation
- posterior glenohumeral (PG) mobilization + thoracic manipulation (Experimental): The group will receive a posterior glide mobilization at session #1, and a thoracic manipulation followed by posterior glide mobilization at session #2.
  Interventions: Other: posterior glide mobilization; Other: thoracic manipulation

INTERVENTIONS:
Other: posterior glide mobilization — The participant will be positioned supine on a plinth, with their scapula stabilized against a firm wedge on the table, and the shoulder joint in the resting position (approx. 55 degrees abduction, 30 degrees horizontal adduction, and slight external rotation). With the extremity held in the same position, the researcher will then apply a grade III (into tissue stretch) PG mobilization. This will consist of five 30-second bouts of sustained gr III posterior glide mobilizations.
  Arms: posterior glenohumeral (PG) mobilization + thoracic manipulation
Other: Sleeper stretch — All participants randomized to the stretching group will perform five 30-second holds of the sleeper stretch. This is performed by lying on the side to be stretched, elevating the upper arm to 90° on the support surface with the elbow bent 90°, then passively internally rotating the shoulder with force provided by with the opposite arm.
  Arms: sleeper stretch + thoracic manipulation
Other: thoracic manipulation — Individuals will then undergo a single supine grade V thrust manipulation. All manipulations will take place at the T3-4 segment. If a cavitation ("pop") is not heard or felt by either the subject or examiner, a second thrust will be performed.

SUMMARY:
Interventions including glenohumeral mobilization, sleeper stretches, and thoracic manipulation have been proposed for individuals with loss of shoulder range of motion (ROM). However, the effect of these interventions on shoulder ROM, joint translation, and muscular activity have not been studied in combination.

DETAILED DESCRIPTION:
Forty individuals with a loss of internal rotation (IR) ROM will be recruited and randomized to one of two interventions at the first session: either posterior glenohumeral mobilization or internal rotation "sleeper" stretching. At the second visit, all participants will undergo a thoracic manipulation (T3-4 segment) followed by a repeat of either the sleeper stretch or glenohumeral mobilization.

ELIGIBILITY:
Inclusion Criteria:

* loss of IR of 15 degrees of greater compared to contralateral shoulder

Exclusion Criteria:

* currently neck/upper back pain,
* history of spinal fractures,
* numbness/altered sensation of the arms or legs,
* whiplash injury within the prior 6 weeks,
* infections of the spine,
* currently pregnant/possibly pregnant,
* known osteoporosis,
* Rheumatoid arthritis,
* previous spine surgery,
* currently receiving Workman's Compensation,
* any pending litigation regarding a neck or shoulder injury,
* history of oral corticosteroids in the prior 6 months,
* history of shoulder fractures,
* Current treatment for cancer,
* Prior history of cancer involving the spine/shoulder,
* any history of coagulation disorders.
* Individuals with a history of shoulder surgery will reviewed on a case by case basis.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-31 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in shoulder IR ROM | Pre intervention to immediate (within 5 minutes) post intervention
  Shoulder IR ROM measured with a goniometer
Change in posterior shoulder translation (mm) | Pre intervention to immediate (within 5 minutes) post intervention
  maximum posterior translation of the humeral head assessed with ultrasound imaging (mm)
Change in infraspinatus electromyographic activity (%MVIC) | Pre intervention to immediate (within 5 minutes) post intervention
  activity of the infraspinatus muscle during posterior translation, assessed as a percentage of the maximal voluntary isometric contraction (MVIC)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Swanson, PT, DSc, Principal Investigator — University of Hartford
Locations (1):
- University of Hartford, West Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No